CLINICAL TRIAL: NCT04656236
Title: Metabolic Effects of Exogenous 3-hydroxybutyrate in Patients With Type 1 Diabetes and Healthy Controls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1-10-72-251-20
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2021-12

CONDITIONS: Type 1 Diabetes Mellitus; Diabetic Ketoacidosis
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Ketoacidosis | interventions — 3-Hydroxybutyric Acid

STUDY DESIGN:
Intervention Model Description: Crossover design in 2 different groups, patients with type 1 diabetes and healthy controls.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 3 hours of continuously intravenous infusion of 3-hydroxybutyrate.
  Interventions: Biological: 3-hydroxybutyrate
- Control (Placebo Comparator): 3 hours of continuously intravenous infusion of saline (NaCl).
  Interventions: Biological: 3-hydroxybutyrate

INTERVENTIONS:
Biological: 3-hydroxybutyrate — 3-hydroxybutyrate is a metabolite, produced in the human body.

SUMMARY:
The main objective of this clinical trial is to study the metabolic effects of intravenous infusion of the ketone body, 3-hydroxybutyrate (3-OHB), in patients with type 1 diabetes and healthy control subjects. Moreover, the investigators plan to examine regulatory mechanisms of 3-OHB that may be related to diabetic ketoacidosis.

The hypotheses are:

1. 3-OHB related inhibition of lipolysis is impaired in patients with type 1 diabetes.
2. Intravenous infusion of 3-OHB affects signaling pathways involved in the metabolic regulation in patients with type 1 diabetes and healthy controls.
3. 3-OHB infusion improves cardiac function in patients with type 1 diabetes and healthy controls.

The effects of 3-OHB will be investigated by isotopic tracers examinations, fat and muscle biopsies and blood samples. To evaluate effects on cardiac function echocardiography will be performed.

ELIGIBILITY:
Patients with type 1 diabetes:

Inclusion Criteria:

* Type 1 diabetes diagnosis
* C-peptide negative
* 19 < BMI < 26
* written consent

Exclusion Criteria:

* Severe comorbidity
* Regular medication apart from insulin (except over-the-counter medicines)
* Use of long acting insulin analogues, that work > 24 hours, e.g. Tresiba
* PI finds the patient not fit (e.g. mental illness, too nervous, unacceptable screening blood tests or other).

Healthy control subjects:

Inclusion Criteria:

* 19 < BMI < 26
* written consent

Exclusion Criteria:

* Chronic disease
* Regular medication (except over-the-counter medicines)
* PI finds the patient not fit (e.g. mental illness, too nervous, unacceptable screening blood tests or other).

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Differences in lipolysis rate | After 3 hours of interventions
  Measured as differences in palmitate flux

SECONDARY OUTCOMES:
Changes in protein metabolism | After 3 hours of interventions
  Measured as differences in forearm and whole body tracer kinetics
Changes in glucose kinetics | After 3 hours of interventions
  Measured by glucose tracer.
Cardiac function | After 2-3 hours of interventions
  Changes in cardiac output and left ventricular ejection fraction measured by echocardiography
Changes in signaling in muscle and adipose tissue | After 1,5-3 hours of interventions
  Western blot examinations of muscle and adipose tissue biopsies
Differences in circulating concentrations of 3-hydroxybutyrate, glucose, free fatty acids, insulin, glucagon and C-peptide | During the 3 hours intervention period
  Blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Niels Møller, Professor, Study Director — Department of Endocrinology and Steno Diabetes Center Aarhus, Aarhus University Hospital; Maj Bangshaab, MD, Principal Investigator — Steno Diabetes Center Aarhus and Aarhus University
Locations (1):
- Steno diabetes center Aarhus, Aarhus, Denmark

REFERENCES:
- [Derived] Bangshaab M, Svart MV, Rittig N, Pedersen MGB, Voigt J, Jessen N, Moller N. Metabolic effects of 3-hydroxybutyrate infusion in individuals with type 1 diabetes compared with healthy control participants: a randomised crossover trial showing intact feedback suppression of lipolysis. Diabetologia. 2025 Jul;68(7):1390-1402. doi: 10.1007/s00125-025-06423-5. Epub 2025 Apr 10. PMID 40210728